CLINICAL TRIAL: NCT04053296
Title: Morbidity and Outcomes of Pregnant Women With Pulmonary Arterial Hypertension During Different Pregnancies
Brief Title: Long-term Outcomes of Pregnant Women With PAH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: outcomes of PAH
Record Dates: First submitted 2019-08-09; First posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The first pregnancy with PAH group
  Interventions: Other: Observational study
- The second pregnancy with PAH group
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — We follow up the results of patients.

SUMMARY:
The investigators intend to explore the characteristics and outcomes of pregnant women with PAH during different pregnancies and to provide applicable evidence for clinical practice.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a fatal disease with progressive vascular resistance that leads to the loss of right heart function. Avoiding pregnancy is essential for PAH women. In recent years, maternal mortality in pregnant women with PAH has decreased mostly due to emerging advanced therapies for PAH and the progress in high-risk pregnancy management. Nevertheless, the maternal death rate in parturients with PAH remains high; therefore, contraception is still recommended for women diagnosed with PAH. However, some women develop this condition during pregnancy. With the two-child policy, families in China are allowed to have a second child. As a result, the number of PAH diagnoses during pregnancy may increase with the general increase in the number of pregnant women. Additionally, some patients develop PAH only during their second pregnancy. In order to investigate the incidence and clinical characteristics of pregnant women diagnosed with PAH during different pregnancies, this observational study aimed to analyze perinatal and pregnancy clinical data, to compare the perinatal status and maternal and infant outcomes of the first and second pregnancies complicated with PAH, establishing a clinical basis for the prenatal consultation, diagnosis, and treatment of pregnant women with PAH.

ELIGIBILITY:
Inclusion Criteria:

PAH was screened by Doppler echocardiography first. Echocardiographic criteria for the diagnosis of PAH included tricuspid regurgitation velocity >2.8 m/sec, with extra more than one additional echocardiographic sign

Exclusion Criteria:

Cases of PH diagnosed before pregnancy, secondary to chronic lung disease, and left heart disease, as well as right ventricular outflow tract obstruction and congenital pulmonary stenosis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The first pregnancy group was composed of patients diagnosed with PAH in their first pregnancy. Patients in the second pregnancy group were diagnosed with PAH during their second pregnancy but normal in their first pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | 10 year
  The patient die at any time.

CONTACTS AND LOCATIONS:
Overall Officials: Jieyan Shen, PhD, Study Chair — Shanghai Jiao Tong University School of Medicine Affiliated Renji Hospital
Locations (1):
- Renji Hospital, Shanghai, China